CLINICAL TRIAL: NCT05498649
Title: Performance of Dailies Total1® Contact Lenses for Astigmatism in Symptomatic Habitual Reusable Toric Lens Wearers
Status: Completed | Type: Observational
Sponsor: Keith Wan (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor-Investigator, Keith Wan, Optometrist, Scripps Poway Eyecare and Optometry
Organization: Scripps Poway Eyecare and Optometry (Other)
Other Study IDs: KW-22-001
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Bilateral use of DT1fA contact lenses: DT1fA contact lenses
  Interventions: Device: DT1fA

INTERVENTIONS:
Device: DT1fA — DT1fA contact lenses

SUMMARY:
To subjectively evaluate Dailies Total1® contact lenses for astigmatism (DT1fA) performance compared to other common weekly/monthly contact lenses in symptomatic patients.

DETAILED DESCRIPTION:
This study is a single site, prospective, subject-masked, observational study of the subjective performance of DT1fA in symptomatic patients. Subjects will be assessed at a screening visit, and 2 follow-up visits. Clinical evaluations will include measurement of visual acuity, manifest refraction, and patient questionnaires.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

Inclusion Criteria:

* Willing and able to provide informed consent
* Adult (18-38 years of age)
* Adapted and optimized current reusable soft toric lens wearer who has at least 3 months of wearing experience, and typically wears lenses every day, or at least 5 days per week, ≥10 hours per day
* Prescription needs with sphere and cylinder values that can be appropriately fit with current available parameters in the Dailies Total1® Contact lenses for Astigmatism product line
* Vision correctable to 20/25 Snellen (0.1 logMAR) or better in each eye at 6m
* Willing to wear lenses every day or at least 5 days per week, 10 or more hours per day and attend all study visits and follow instructions
* CLDEQ-8 minimum score of 12

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Ocular anterior segment infection, inflammation, abnormality, or active disease including diagnosed dry eye, that would contraindicate contact lens wear
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the Investigator
* Monocular (only 1 eye with functional vision) or fit with only 1 lens
* Fitted with monovision
* Prior Refractive Surgery
* History of herpetic keratitis, ocular surgery, or irregular cornea
* Pregnant or lactating

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Ages: 18 Years to 38 Years | Sex: All
Age Groups: Adult
Study Population: Eligible participants will be 18-38 years of age who are current and appropriate candidates for contact lens wear.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wan, OD, Principal Investigator — Scripps Poway Eyecare & Optometry
Locations (1):
- Scripps Poway Eyecare & Optometry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral Use of DT1fA Contact Lenses
Started | 86
Completed | 85
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bilateral Use of DT1fA Contact Lenses
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score
Description: A series of 8 questions that ask participants to rate eye discomfort, eye dryness, and blurry vision on a frequency scale (0 Never, 1 Rarely, 2 Sometimes, 3 Frequently, 4 Constantly) and an intensity scale (0 Never, 1 not intense to 5 Very Intense). Scores on individual questions are added together to determine a total score. Higher values indicate worse outcomes. The minimum score is 1 and the maximum score is 37.
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Habitual Lens: New habitual toric lenses with an optimized prescription
- Delefilcon A: Refit with delefilcon A for astigmatism
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
score on a scale | 16.8 (8.1) | 12.4 (7.5)

2. Other Pre Specified Outcome: The Percentage of Participants That Reported Little to no Intensity of Eye Discomfort at Baseline and 2 Weeks of DT1fA Wear for End of Day (EOD)
Description: Participants were asked to rate end of day discomfort intensity (0 Never, 1 not intense to 5 Very Intense). Higher values indicate worse outcomes.
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Population: Percentage that reported little to no intensity of eye discomfort (responding 0, 1, or 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
Participants | 67 | 44

3. Other Pre Specified Outcome: The Percentage of Participants That Reported Little to no Intensity of Eye Dryness at Baseline and 2 Weeks of DT1fA Wear for End of Day (EOD)
Description: Participants were asked to rate end of day dryness intensity (0 Never, 1 not intense to 5 Very Intense). Higher values indicate worse outcomes.
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Population: Percentage that reported little to no intensity of dryness (responding 0, 1, or 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
Participants | 66 | 43

4. Other Pre Specified Outcome: The Percentage of Participants That Reported Little to no Noticeable Change Between Clear to Blurry or Foggy Vision at Baseline and 2 Weeks of DT1fA Wear for End of Day (EOD)
Description: Participants were asked to rate noticeable change between clear to blurry or foggy vision (0 Never, 1 not intense to 5 Very Intense). Higher values indicate worse outcomes.
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Population: Percentage that reported little to no noticeable change between clear to blurry or foggy vision (responding 0, 1, or 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
Participants | 55 | 46

5. Other Pre Specified Outcome: Hours of Comfortable Wear
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
hours | 9.0 (4.8) | 8.0 (4.1)

6. Other Pre Specified Outcome: Vision Stability
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Binocular Contact Lens Corrected Visual Acuity at Distance (6m)
Time Frame: Two to four weeks after fit with optimized prescription (Habitual lens) or two weeks after refit (Delefilcon A)
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Habitual Lens | Delefilcon A
Number analyzed (Participants) | 85 | 85
logMAR | 0.00 (0.09) | 0.05 (0.12)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Bilateral Use of DT1fA Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT05498649/Prot_SAP_000.pdf